CLINICAL TRIAL: NCT01511055
Title: Phase II, Prospective, Non-Randomized Trial Investigating the Intra-Operative Detection of Occult Ovarian Carcinoma Using a Folate-Alpha Receptor Specific Fluorescent Ligand
Brief Title: Intra-op Detection of Occult Ovarian Carcinoma Using a Folate-Alpha Receptor Specific Fluorescent Ligand
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual temporarily suspended, followed by study closure due to technical problems with investigational camera.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sean C Dowdy, MD, Associate Professor - Obstetrics and Gynecology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-002980
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Folate-FITC (Experimental)
  Interventions: Drug: EC-17

INTERVENTIONS:
Drug: EC-17 — One-time dose of Folate-FITC (EC-17), 0.1mg/kg IV 2-3 hours prior to surgery.
  Other Names: Folate-FITC

SUMMARY:
Prognosis for many carcinomas, including ovarian carcinoma, is dependent on a complete surgical resection, also known as a R0 resection. At present, the ability to perform a complete resection with negative margins is limited by the surgeon's ability to palpate and visualize the tumor and its margins. Therefore, in order to reduce operative morbidity and costs while maintaining or improving surgical and oncologic outcomes, the investigators must develop technologies that improve visualization of the primary tumor and occult metastases, real time, during surgery. Recent research has demonstrated that the use of fluorescent probes that recognize cancer specific antigens can be used for this purpose when visualized using a prototype near-infrared multispectral imaging system.

This investigation will determine if folate-FITC, a fluorescent probe that recognizes the folate receptor (present in > 90% of ovarian cancers) can facilitate surgical resection and detect tumor nodules not visible to the naked eye.

ELIGIBILITY:
Inclusion Criteria:

Women who are:

* Diagnosed with or at high clinical suspicion of primary ovarian cancer by either radiologic imaging or physical examination or biopsy or serum tumor markers
* Scheduled to undergo surgical cytoreduction via laparotomy
* At least 18 years of age
* Capable and willing to provide informed consent

Exclusion Criteria:

Women with:

* Known sarcomatous histologies
* Recurrent ovarian cancer
* Planned surgical approach via laparoscopy or robotic surgery
* A history of anaphylactic reactions to Folate-FITC or insects
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean C Dowdy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Folate-FITC
Started | 27
Completed | 21
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Folate-FITC
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  Age 40-49 | 3
  Age 50-59 | 6
  Age 60-69 | 9
  Age 70-79 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Intra-operative Imaging Using Folate-FITC for Identification of Ovarian Cancer Metastatic to the Peritoneum and Lymph Nodes
Description: A maximum of 5 nodules less than 1cm in size will be identified in each patient with the naked eye and then visualized with the camera. The nodules will be biopsied after determining if they are fluorescent positive or negative (F+ or F-), and examined microscopically to confirm if carcinoma is present. Up to 5 F+ lesions that were not identified with the naked eye will also be biopsied and examined microscopically to determine if carcinoma is present. These data will establish the sensitivity and specificity of this technique using microscopic analysis as the gold standard.
Time Frame: 1 week
Population: The investigational camera was instrumental for collecting data for this study. Due to technical problems with the camera from the onset of the study, the study was terminated and no data was able to be collected or analyzed.
Arm/Group | Folate-FITC
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Grade 4 or Higher Adverse Events Following a One-time Dose of Folate-FITC (EC-17).
Description: Study participants will be followed and all adverse events will be captured for the duration of hospitalization following administration of investigational product, up to a maximum of 7 days following IP administration and surgical procedure. Adverse Events will be classified as: grade 1=Mild, grade 2=Moderate, grade 3=Severe, grade 4=Life-threatening/disabling, grade 5 =Death. Significant is defined as adverse events grade 4 or higher.
Time Frame: Duration of hospitalization with a maximum of 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Folate-FITC
Number analyzed (Participants) | 27
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the period from the initiation of any study procedures to the end of the study treatment follow-up, approximately one week
Arm/Group | Folate-FITC
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 15/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folate-FITC (N=27)
Sneezing, spontaneous onset (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tingling sensation in mouth, palate and molars (Gastrointestinal disorders) | 3 (3)
Mild facial flusing (Vascular disorders) | 2 (2)
Sinus pressure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Plugged ears (Ear and labyrinth disorders) | 1 (1)
Strong taste in mouth (Gastrointestinal disorders) | 1 (1)
Cirumoral and Nasal Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The investigational camera was instrumental for collecting data for this study. Due to technical problems with the camera from the onset of the study, the study was terminated and no data was able to be collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes